CLINICAL TRIAL: NCT00325611
Title: A Multi-Site Replication of an Inpatient Palliative Care Program
Brief Title: Multidisciplinary Inpatient Palliative Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Garfield Memorial Fund (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CO-02GGade-01 - H; NW-02RRich-01
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2006-05

CONDITIONS: Cerebrovascular Accident; Cancer; Coronary Arteriosclerosis; Heart Failure, Congestive; Diabetes Mellitus; Acquired Immunodeficiency Syndrome; Failure to Thrive; Pulmonary Disease, Chronic Obstructive; Dementia; Kidney Failure, Chronic; Pneumonia; Liver Failure; Renal Failure; Respiratory Failure; Stroke
Keywords: Palliative care; End of life care
MeSH Terms: conditions — Stroke; Neoplasms; Coronary Artery Disease; Heart Failure; Diabetes Mellitus; Acquired Immunodeficiency Syndrome; Failure to Thrive; Pulmonary Disease, Chronic Obstructive; Dementia; Kidney Failure, Chronic; Pneumonia; Liver Failure; Renal Insufficiency; Respiratory Insufficiency

INTERVENTIONS:
Behavioral: Multidisciplinary palliative care team met with patient

SUMMARY:
Palliative care is believed to improve care of patients with life-limiting illnesses. This study evaluated the impact of a multi-center randomized trial of a palliative care team intervention on the quality and cost of care of hospitalized patients. Study subjects were randomized to intervention or usual care. At study end, patients receiving the palliative care intervention reported greater patient satisfaction with their care. Intervention patients also had significantly fewer ICU admissions and lower total costs for care 6 months past their hospitalization. Intervention patients completed more advance directives and had longer hospice stays.

DETAILED DESCRIPTION:
The Inpatient Palliative Care Service (IPCS) was implemented at three Kaiser-Permanente sites: Colorado, Portland and San Francisco. The service consisted of a physician, nurse, social worker, and spiritual counselor who worked with the study subjects randomized to receive the intervention. The intervention included symptom control, emotional and spiritual support, advance care and post-discharge care planning, There were no differences in symptom control or emotional support but IPCS patient reported better spiritual support compared to usual care patients. IPCS patients also reported greater satisfaction with their hospital care experience and better communication with their providers. Both IPCS and usual care patients reported improved quality of life during their enrollment hospital stay. IPCS patients completed more advance directives. IPCS patients had more home health visits than usual care patients but significantly fewer ICU admissions. IPCS patients had significantly lower hospital costs and higher pharmacy costs, than the usual care patients. IPCS patients had significantly lower (p= .001) total health services costs (a cost savings of $64.90 per patient per day) compared to usual care patients. This translated to an average total cost savings of $3,185 per enrolled patient. IPCS patients had a significantly longer average hospice length of stay. There were no differences between IPC and usual care patients in the proportion admitted to hospice, time to hospice admission, the average length of survival, or proportion of those who survived to 6 months.

Conclusion: IPCS resulted in better spiritual support, a better hospital care experience, better communication with their providers, increased completion of advance directives, fewer ICU admissions, longer hospice stays and reduced overall health care costs.

ELIGIBILITY:
Inclusion Criteria:

Adults 18 years and older

-admitted to acute inpatient care who had: (1) a medical diagnosis which was life-threatening, and (2) whose attending physician indicated they "would not be surprised if the patient died within one year".

Exclusion Criteria:

* 1) they had impaired cognitive status and no caregiver was available to provide consent, (2) were currently enrolled in hospice or other studies involving palliative care, (3) the attending physician did not approve study participation, or (4) their medical condition impaired participation (actively dying, too ill to participate) and no family member was available to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2002-04; Study Completion 2004-07

PRIMARY OUTCOMES:
Quality and cost of care

SECONDARY OUTCOMES:
Greater patient satisfaction
Lower ICU admissions
Lower total costs 6 months past hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid M Venohr, RN, PhD, Study Director — Kaiser Permanente; Douglas A Conner, PhD, Principal Investigator — Kaiser Permanente Northwest Region; Marcia Liberson, MSW,MPH, Principal Investigator — Kaiser-Permanente Northwest Region
Locations (1):
- Kaiser Permanente of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Result] Conner D. Differences in survival, hospice admission, and hospice length of stay for patients randomized to either an inpatient palliative care team intervention or to usual care. Poster presentation at the American Geriatrics Society Annual Meeting. May 2005.
- [Result] Conner D, McGrady K, Richardson R, Beane J. Predictors of Hospice Admission and Length of Stay from a Randomized Control Trial of an Inpatient Palliative Care Service. Paper presentation at the American Academy of Hospice and Palliative Medicine annual meeting. February 2006, Nashville, TN.
- [Result] McGrady K, Conner D, Richardson R, Beane J, Connors L, Rastrelli A, Collins T. Influence of an Inpatient Palliative Care Team on Service Utilization and Costs. Paper presentation at the American Academy of Hospice and Palliative Medicine annual meeting. February 2006, Nashville, TN.
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Gade G, Venohr I, Conner D, McGrady K, Beane J, Richardson RH, Williams MP, Liberson M, Blum M, Della Penna R. Impact of an inpatient palliative care team: a randomized control trial. J Palliat Med. 2008 Mar;11(2):180-90. doi: 10.1089/jpm.2007.0055. PMID 18333732